CLINICAL TRIAL: NCT05548595
Title: A Prospective, Randomized, Proof of Concept Study to Evaluate the Impact of a Nutritional Product on Cognition in Healthy Teenagers
Brief Title: A Study to Evaluate the Impact of a Nutritional Product on Cognition in Healthy Teenagers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hong Kong Prospect Group Co. Limited (Industry)
Collaborators: Nutrasource Pharmaceutical and Nutraceutical Services, Inc. (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: H02-21-01-T0018
Record Dates: First submitted 2022-09-17; First posted 2022-09-21 (Actual); Last update posted 2022-09-21 (Actual); Status verified 2022-09

CONDITIONS: Healthy

STUDY DESIGN:
Intervention Model Description: Randomization at 1:1 ratio for active or placebo
Who Masked: Participant, Investigator
Masking Description: Double blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Investigational (Experimental): Active ingredients (per tablet):
  • NeumentixTM Phenolic
  Complex K110-42:
  * 450 mg Spearmint extract (Mentha spicata)
  * 100 mg Alpha-Glyceryl Phosphoryl Choline
  * 50 mg Phosphatidylserine (Sharp PS®)
  * 10 mg Pyrroloquinoline quinone
  Inactive ingredients (per tablet):
  * Microcrystalline cellulose
  * Maltodextrin
  * Hardened rapeseed fat
  * Magnesium salts from fatty acids (palm oil free)
  * Silicon dioxide
  * Glycerin
  * Hydroxypropyl methylcellulose
  Interventions: Dietary Supplement: Investigational
- Placebo (Placebo Comparator): Active ingredients (per tablet):
  N/A
  Inactive ingredients (per tablet):
  * Lactose monohydrate
  * Magnesium stearate
  * Microcrystalline cellulose
  Interventions: Other: Placebo

INTERVENTIONS:
Dietary Supplement: Investigational — 2 tablets are taken with water around the same time every day, ideally after a meal
  Other Names: BDF Mega Brain Boost
  Arms: Investigational
Other: Placebo — 2 tablets are taken with water around the same time every day, ideally after a meal
  Arms: Placebo

SUMMARY:
Nutritional products such as spearmint extract, alpha-glyceryl phosphoryl choline and phosphatidylserine may have anti-oxidative and anti-inflammatory effect that may be effective in improving cognition. This study aims to evaluate the impact of a nutritional product on cognition in healthy teenagers.

DETAILED DESCRIPTION:
There is a growing interest in the nootropic properties of nutritional supplements, especially for improving cognitive processes such as attention, perception, evaluation, and working memory. Spearmint extract, alpha-glyceryl phosphoryl choline, and pyrroloquinoline quinone have antioxidative properties that may contribute to cognitive function, and spearmint extract has demonstrated attention-enhancing effects in young adults and memory-improving effects in elderly population. Phosphatidylserine is a phospholipid found abundantly in the brain that has also been evidenced to be effective in improving cognition.

This randomized, double-blind study will be conducted to determine whether a nutritional supplement containing spearmint extract, phosphatidylserine, alpha-glyceryl phosphoryl choline, and pyrroloquinoline quinone ("Brain Doctors Formula Mega Brain Boost") is safe and effective in improving cognitive function in healthy participants aged 12 to 18 years.

ELIGIBILITY:
Inclusion Criteria:

1. Middle, high school, or college students who are 12 to 18 years of age (inclusive).
2. In good general health (no active or uncontrolled diseases, infections, or conditions) and able to swallow the study products (tablets).
3. Have normal (or acceptable to the investigator) vital signs (blood pressure and heart rate) at screening.
4. Individuals of childbearing potential must practice a medically acceptable form of birth control for a certain timeframe prior to the first dose of study product and throughout the study, including:

   1. use for at least 3 months prior to the first dose of study product: hormonal contraceptives including oral contraceptives, hormone birth control patch (e.g., Ortho Evra), vaginal contraceptive ring (e.g., NuvaRing), injectable contraceptives (e.g., Depo-Provera, Lunelle), or hormone implant (e.g., Norplant System); or
   2. use for at least 1 month prior to the first dose of study product: double-barrier method, intrauterine devices or
   3. vasectomy of partner at least 6 months prior to the first dose of study product Individuals of the potential to get others pregnant must use condoms or other medically acceptable methods to prevent pregnancy throughout the study.
5. Agree to refrain from treatments listed in protocol in the defined timeframe.
6. Participant and participant's legally authorized representative (LAR, if applicable) are willing and able to agree to the requirements and restrictions of this study, be willing to give voluntary consent and assent, be able to understand and perform the assessments, carry out all study-related procedures, communicate effectively with the study staff, and agree to allow evaluations related to cognitive function.

Exclusion Criteria:

1. Female or transgendered male participants who are lactating, pregnant or planning to become pregnant during the study.
2. History of diagnosis of depression, other psychiatric disorders (e.g., attention deficit hyperactivity disorder [ADHD]), or any related condition within the past five years.
3. History of heart disease/cardiovascular disease, uncontrolled hypertension (i.e., ≥130 mmHg systolic and/or ≥80 mmHg diastolic), kidney disease (dialysis or renal failure), hepatic impairment, Type I or Type II diabetes, unstable thyroid disease, immune disorder (i.e., HIV/AIDS), or cancer (except localized skin cancer without metastases or in situ cervical cancer) within 5 years prior to screening visit.
4. Have a known sensitivity, intolerability, or allergy to any of the study products or their excipients.
5. Use of concomitant treatments listed in protocol within the defined timeframe.
6. Any condition or abnormality that, in the opinion of the investigator, would compromise the safety of the participant or the quality of the study data.
7. History of alcohol or substance abuse in the 12 months prior to screening.
8. Receipt or use of test product(s) in another research study within 28 days prior to baseline (Visit 2) or longer if the previous test product is deemed by the investigator to have lasting effects that might influence the eligibility criteria or outcomes of current study.
9. Siblings or family members living at the same address if there is already a participant from the same family/address.
10. Any other active or unstable medical conditions or use of medications/supplements/ therapies that, in the opinion of the investigator, may adversely affect the participant's ability to complete the study or its measures or pose a significant risk to the participant.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 22 (Actual)
Dates: Start 2022-01-29 (Actual); Primary Completion 2022-04-04 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
To determine the impact of test product on the executive cognitive function in healthy adolescents within the group and when compared to the placebo | after 3 and 6 weeks
  Change from baseline in national institute of health (NIH) Toolbox Dimension Change Card Test (aged 12+ version) after 3 and 6 weeks. Dimensional Change Card Sort Test is a measure of cognitive flexibility. The scoring range is provided as an age-corrected normative score. A score of 100 indicates performance that is at the national average for the participant's age. A score of 115 or 85 would indicate that the participant's performance is 1 SD above or below the national average, respectively, when compared with like-aged participants
To determine the impact of test product on the attention and executive cognitive function in healthy adolescents within the group and when compared to the placebo | after 3 and 6 weeks
  Change from baseline in NIH Toolbox Flanker Inhibitory Control and Attention Test (12+) after 3 and 6 weeks. The Flanker task measures both attention and inhibitory control. A score of 100 indicates performance that is at the national average for the participant's age. A score of 115 or 85 would indicate that the participant's performance is 1 SD above or below the national average, respectively, when compared with like-aged participants
To determine the impact of test product on the cognitive processing speed of healthy adolescents within the group and when compared to the placebo | after 3 and 6 weeks
  Change from baseline in NIH Toolbox Pattern Comparison Speed Test after 3 and 6 weeks. This test measures speed of cognitive processing. A score of 100 indicates performance that is at the national average for the participant's age. A score of 115 or 85 would indicate that the participant's performance is 1 SD above or below the national average, respectively, when compared with like-aged participants
To determine the impact of test product on the working memory of healthy adolescents within the group and when compared to the placebo | after 3 and 6 weeks
  Change from baseline in the Symmetry Span Task after 3 and 6 weeks. The symmetry span task is a measure of working memory capacity. Scores on the task range from 0-42 with higher scores representing greater working memory capacity
To determine the impact of test product on self reported mind wandering of healthy adolescents within the group and when compared to the placebo | after 3 and 6 weeks
  Change from Week 1 in the self assessment of mind wandering, as captured in a study daily diary, after 3 and 6 weeks by using the The Mind Wandering Questionnaire. The Mind Wandering Questionnaire is a retrospective measure of mind wandering in a everyday life. A scoring range is between 1-6. Higher scores on this scale represent greater levels of mind wandering experienced
To assess the safety and tolerability of the test product in healthy adolescents | 6 weeks
  Counting the number of adverse events over the study period
To assess the safety and tolerability of the test product in healthy adolescents | 6 weeks
  Assessing the type of adverse events (non serious or serious) over the study period
To assess the safety and tolerability of the test product in healthy adolescents | 6 weeks
  Assessing the severity of adverse events (mild, moderate, severe) over the study period

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Tartar, Ph.D., Principal Investigator — Nova Southeastern University
Locations (1):
- Nova Southeastern University, Fort Lauderdale, Florida, United States

IPD SHARING:
Plan to Share IPD: No